CLINICAL TRIAL: NCT06416631
Title: Artificial Intelligence Versus Manual Planning in Patients Undergoing Robot-assisted Pedicle Screw Internal Fixation: a Prospective Controlled Study
Brief Title: Artificial Intelligence Versus Maunal Planning in Robot Assisted Spinal Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI-RASS
Record Dates: First submitted 2024-04-27; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- artificial intelligence planning group (Experimental)
  Interventions: Procedure: artificial intelligence based screw planning
- manual planning group (Placebo Comparator)
  Interventions: Procedure: manually screw planning

INTERVENTIONS:
Procedure: artificial intelligence based screw planning — artificial intelligence technology helps to plan screws in robot assisted spinal surgery
  Arms: artificial intelligence planning group
Procedure: manually screw planning — the screw trajcetories are manually planned
  Arms: manual planning group

SUMMARY:
The goal of this clinical trial is to learn if the artificial intelligence technology helps to improve the efficiency in robot assited spinal surgery. The main questions it aims to answer are:

Does the AI technology shorter the mannual planning time of screw trajectories？ Does the AI technology affect the surgical accuracy？ Researchers will compare the artificial intelligence technology to the conventional mannual planning in robotic surgery.

Participants who met inclusion criteria and do not have any exclusion criterion will be randomized to artificial intelligence or mannual planning group.

DETAILED DESCRIPTION:
Study design:

multicenter, non-inferiority, open-label, randomized controlled trial in patients undergoing robotic spinal surgery.

Monitoring:

Monitoring of patient's safety and effectiveness data is performed by a designated independent Data Safety and Monitoring Board (DSMB). The DSMB watches over the ethics of conducting the study in accordance with the Declaration of Helsinki.

Sample Size Calculation:

Group size calculation is focused on demonstrating non-inferiority. Assuming that the percentage of clinically acceptable screws would be 90% in the artificial intelligence planning group and 95% in the manual planning group, with a non-inferiority margin of 10% and a one-sided significance level of 2.5%, we calculated that a sample of 79 screws per treatment group would give the trial approximately 95% power to show noninferiority of artificial intelligence planning group to manual planning group with regard to the primary end point.

ELIGIBILITY:
Inclusion Criteria:

* Admission to one of the participating centers；
* Need for and start of robotic spinal surgery
* Patients had complete medical records and imaging data;

Exclusion Criteria:

* Age less than 18 years;
* Patients with severe comorbidities;
* Patients diagnosed with tumor diseases;
* Inability to carry out the intervention (mental of physical conditions that limited participation);
* Patients with morbid obesity (body mass index > 40);
* Missing medical records and imaging data;
* Patients with suspected or confirmed pregnancy;
* Patients participating in another RCT with the same clinical endpoint, or interventions possibly compromising the primary outcome;
* No informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-25 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
The accuracy of screw positioning or placement | 1 month
  according to the Gertzbein and Robbins scale, including grade A (screw was completely within the pedicle), grade B (pedicle cortical breach <2 mm), grade C (pedicle cortical breach <4 mm), grade D (pedicle cortical breach <6 mm), and grade E (pedicle cortical breach >6 mm). Grade A + B were considered clinically acceptable. The percentage of clinically acceptable screws was recorded.

SECONDARY OUTCOMES:
The planning time | 1 day
  Time from start to finish of planning
postoperative complication | 3 month
  Nerve injury, epidural hematoma, and infection